CLINICAL TRIAL: NCT00842049
Title: Lumbar Drainage of Cerebrospinal Fluid in Aneurysmal Subarachnoid Haemorrhage: A Prospective Randomised Controlled Trial
Brief Title: Lumbar Drainage in Subarachnoid Haemorrhage
Acronym: LUMAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/Q1205/170
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid haemorrhage; Aneurysm; Cerebrospinal fluid drainage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm; Cerebrospinal Fluid Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study (Experimental): Insertion of lumbar drain
  Interventions: Device: Lumbar Drain (Medtronic lumbar drainage system)
- Control (Other): Normal clinical management without lumbar drain
  Interventions: Other: No lumbar drain

INTERVENTIONS:
Device: Lumbar Drain (Medtronic lumbar drainage system) — Insertion of lumbar drain to drain cerebrospinal fluid
  Other Names: Medtronic lumbar drainage system
  Arms: Study
Other: No lumbar drain — No lumbar drain
  Arms: Control

SUMMARY:
Subarachnoid haemorrhage affects approximately 8000 people per year in the UK. The average age of a patient with subarachnoid haemorrhage is 50 years, although it is often seen in younger people (25-45 years). Despite modern medicine, the death and disability rate remains high both from the initial bleed and from the associated complications such as vasospasm. This is characterised by neurological impairment seen following the bleed. Despite modern treatment this is still associated with a poor outcome. This has significant implications due to the long term intensive neuro-rehabilitation these patients will require.

A recent study has shown that placing a small drain in the lower back following a subarachnoid haemorrhage may reduce the chance of vasospasm occurring and result in a better outcome. This trial was not optimally performed and so a trial is needed to look at this in more detail. The investigators have set up such a trial in our neurosurgical unit. If the investigators confirm that there is an improvement in patient outcome, it will change our practice in the future.

DETAILED DESCRIPTION:
All patients who present to our department with proven aneurysmal SAH and fit the inclusion criteria (see below) will be approached for inclusion into the trial. Written informed consent will be sought prior to recruitment into the study. Written assent from the patient's relatives will be sought in those cases where neurological impairment prevents written informed consent being obtained from the patient. The patient will subsequently be randomised into the control arm or the study arm of the trial. The control arm consists of normal therapeutic intervention, including external ventricular drainage if required for hydrocephalus. Those randomised to the therapeutic arm will have a lumbar drain inserted and set to drain CSF at 5 ml/hour. This will continue until CSF is no longer blood stained or until day 10 following insertion.

Primary outcome measures:

1. Incidence of delayed ischaemic neurological deficit. This is defined as new neurological deficit and/or impairment of consciousness without other identifiable cause at least three days post haemorrhage.

New impairment of consciousness is defined as a drop in the Glasgow Coma Score of 1 motor point or 2 verbal/eye opening points.

Secondary outcome measures:

1. Modified Rankin Score at day 10 post ictus and at 6 months.
2. Severity of delayed neurological deficit and the development of a complete infarct.
3. Incidence of cerebrospinal fluid infection secondary to lumbar drainage

Special note:

If a patient has presented greater than three days following the initial bleed, any neurological deficit present may be a delayed neurological deficit and thus must be excluded from the trial. Should the lumbar drain fall out prematurely the patient will be asked whether they wish to continue in the study and, if so, the lumbar drain will be reinserted and management will continue as before. Patients showing signs of lumbar drain infection will have the drain removed, a sample of CSF and the drain tip sent to the microbiology laboratory and appropriate antibiotic therapy instituted.

The neurosurgical unit at Leeds General Infirmary treated 313 patients with acute subarachnoid haemorrhage in the three years 1997-2000. Of these 243 patients would have been suitable for this study on the basis of their admission clinical status. The power calculation was derived from the estimate that 40% of patients treated with standard therapy will develop clinical vasospasm. If the retrospective study showed a minimum of 20% improvement in its outcome variables then we expect to see the same improvement. For an 85% power this requires 105 patients in each arm. We expect this to take 3.5 years based on the number of eligible patients that present to our unit with a 60-70% recruitment rate (approximately 30 patients per year per arm).

ELIGIBILITY:
Inclusion Criteria:

1. Aneurysmal subarachnoid haemorrhage.
2. Recruitment prior to day three post-haemorrhage.
3. Written informed consent or relative assent given.
4. WFNS grade 1-3.
5. Fisher grade 2, 3 and 4 (without space occupying haematoma) on initial CT scan.
6. No intraventricular haemorrhage, space occupying haematoma or other contra-indication to lumbar puncture.

Exclusion Criteria:

1. Non-aneurysmal subarachnoid haemorrhage.
2. Delayed presentation / recruitment (after day three post-haemorrhage)
3. Written informed consent or relative assent denied or unobtainable.
4. WFNS grade 4 or 5.
5. Fisher grade 1 on initial CT scan.
6. Intraventricular haematoma obstructing ventricular outflow.
7. Intracranial haematoma with mass effect.
8. Bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2006-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Incidence of delayed ischaemic neurological deficit | Within 21 days of haemorrhagic ictus

SECONDARY OUTCOMES:
Modified Rankin Score | 10 days and 6 months following haemorrhagic ictus
Incidence of cerebrospinal fluid shunting | Within 12 months of haemorrhagic ictus
Incidence of completed infarct secondary to delayed ischaemic neurological deficit | Within 21 days of ictus
Incidence of cerebrospinal fluid infection secondary to lumbar drainage | Within 8 weeks of removal of lumbar drain

CONTACTS AND LOCATIONS:
Overall Officials: Yahia Al-Tamimi, MCChB(Hons), Principal Investigator — Leeds Teaching Hospital NHS Trust; Stuart Ross, FRCS(SN), Study Director — Leeds Teaching Hospital NHS Trust
Locations (1):
- Leeds General Infirmary, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Background] Klimo P Jr, Kestle JR, MacDonald JD, Schmidt RH. Marked reduction of cerebral vasospasm with lumbar drainage of cerebrospinal fluid after subarachnoid hemorrhage. J Neurosurg. 2004 Feb;100(2):215-24. doi: 10.3171/jns.2004.100.2.0215. PMID 15086227
- [Derived] Al-Tamimi YZ, Bhargava D, Feltbower RG, Hall G, Goddard AJ, Quinn AC, Ross SA. Lumbar drainage of cerebrospinal fluid after aneurysmal subarachnoid hemorrhage: a prospective, randomized, controlled trial (LUMAS). Stroke. 2012 Mar;43(3):677-82. doi: 10.1161/STROKEAHA.111.625731. Epub 2012 Jan 26. PMID 22282887